CLINICAL TRIAL: NCT00719082
Title: Fall Prevention:Dynamic Posturographic Measurements in the Geriatric Population
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funding
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal Investigator, Carrick Institute for Graduate Studies
Other Study IDs: CI-IRB-01-7-7-08
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Balance, Falls
Keywords: Human Stability; Geriatric; Posturography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AARP Community: Members of AARP Geriatric Community

SUMMARY:
Falls are the greatest cause of accidental death in the elderly. There is no normative data on large groups of geriatric subjects specific to their stability scores obtained by computerized dynamic posturography (CDP). CDP is the standard test to obtain stability scores and is utilized as the gold standard in posturographic evaluations and fall prevention

Hypotheses:

Human stability can be measured by CDP. Increased stability is associated with a lessor probability of falls. Stability decreases as age increases and a normative data collection of stability scores in the geriatric population will allow and promote clinical applications which can be utilized in fall prevention.

DETAILED DESCRIPTION:
Computerized dynamic posturography outcomes will be obtained on geriatric subjects attending the September, 2008 AARP meeting in Washington, DC. All subjects will be volunteers. The outcome measurement will be obtained using computerized dynamic posturography, a standard diagnostic test of balance function. The subject's balance will be tested using a three-component force platform (CAPS test) under one sensory condition of the modified Clinical Test of Sensory Interaction on Balance (mCTSIB), the eyes closed without perturbation. This condition is chosen as studies have shown it to be the single test that best correlates with balance impairment and falls. The stability score, already used in several studies by other authors will be used as the primary outcome measure in this research. It is defined as 1 minus the ratio between the measured sway during the test (computed as the major axis of a standard 95% confidence ellipse) and the amount of sway a normal subject of the same height as the one being tested should be able to sway before falling (also known as the theoretical maximum sway or the theoretical limit of stability, calculated using a regression formula based on the subject's height developed by NASA in 1962 and commonly used in all posturographic tests). For convenience, the stability score will be expressed as a percentage. Its definition makes it a convenient and easy to understand measure to use as a subject able to stand perfectly still with no sway will have a score of 100%, whereas one that sways as much as the limit of stability will have a score of 0%. During each test, the subject's sway will be determined by the force platform and its related software. The CAPS three-component force platform uses 3 load cells arranged in a triangle to measure the distribution of the vertical ground reaction force on the platform. The analog load cell signals are amplified and simultaneously sampled by the platform electronics using three synchronized individual 24-bit delta-sigma analog to digital converters sampling at 312 kHz and decimating the samples to a data rate of 64 Hz. The use of three A/D converters insures that the signals from the 3 load cells are acquired simultaneously with no timing error. The high sampling rate with the high decimation and low data rate of the sigma-delta converters eliminates aliasing and provides a resolution of about 4 parts per million. The digital load cell data will be then sent via a USB connection to the PC where software uses a calibration matrix determined by the manufacturer to compute the total vertical force and the two horizontal moments acting on the platform. From these data, the software will compute the point of application of the vertical force acting on the platform, commonly referred to as the Center of Pressure (CoP). The location of the CoP coincides in static conditions with the projection of the subject's Center of Mass (CoM) onto the platform, and its movement relates to the movements of the subject's CoM (sway). The determination of the actual sway will require the determination of the instantaneous location of the CoM via the location and inertial properties of each body segment of the specific subject being tested. The CAPS test, like all posturographic equipment, uses the movement of the CoP as an approximation of the sway. Because it is an approximation, and because for kinetic reasons the CoP moves more than the CoM, the 95% confidence interval of the CoP motion will be considered. This will allow the CAPS software to compute the ellipse that represents the location of all of the sway samples collected during the test with 95% confidence. The major axis of this ellipse will represent the maximum sway of the subject in any direction during the test and it will be used to compute the stability score. To assess the accuracy and resolution of the measurement chain, calibrated weights of 75 kg and 100 kg will be positioned in the center of the force platform (as if it were a subject) and 20 sec acquisitions will be performed: The accuracy of the weight must fall within the instrument's factory specifications (+2N). Therefore the accuracy for the position claimed by the manufacturer of +1 mm for a weight of 75 kg will be accepted as correct as it determination would have required specialized equipment and software available only to the manufacturer. It should be noted that the overall accuracy of the position of the CoP given by the instrument will not be relevant in this study as the motion of the CoP will determine the sway. The sway measurement error will be estimated considering the fact that during the test at both weights the dead weight will not move, but the measurement chain will indicate a ''sway'' of less then 0.05 mm (measurement noise), therefore the resolution of the measurement chain and the sway measurement error will be considered to be 0.05 mm. To verify the repeatability of the measurement chain, the same type of tests will be repeated two times. The authors have obtained similar results (within the specified accuracy and resolution) in another study. Given the sway measurement error, the measurement error in the stability score will be determined. From the definition of the stability score it is clear that the least the theoretical limit of stability, the more pronounced the effect of the sway measurement error will be. As the theoretical limit of stability is computed by using the formula 0.556height626sin(6.258), the shorter the subject, the more the stability score is sensitive to the measurement errors. To estimate the stability score measurement error a subject's height of 1.6 m will be considered. Such a subject would have a theoretical limit of stability of 191.6 mm. For such a subject, a sway measurement error of 0.05 mm means a stability score measurement error of 0.05/191.6 or, if the score is expressed in percentage, of 0.026%. Thus, any changes in the stability score greater than that are a consequence of the subject's sway and not of measurement errors. A CAPS sit to stand test in which the subject will be asked to stand on the force platform from a sitting position followed by a posturography test in the eyes closed stance will be obtained on all subjects. Subjects will be instructed that they will sit on a chair and then stand up without using their hands or a structure for support. They then wil be instructed to stand on a computerized force plate platform without pertubation and close their eyes while data is obtained from the computerized force plate. The subjects will be given practice sessions so that they will be familiar with the test prior to the collection of data. The CAPS testing, including the sit to stand and the eyes closed standing test occurs over 90 sec. We will divide the degree of sway observed during the first half of the eyes closed standing test (10 seconds) and the second half of the eyes closed standing test (10 seconds)and obtain ratios. If a subjects sway increases in the second half of the test in reference to the first half we will call this a fatigability ratio. When individuals demonstrate less sway in the second half of the test we will call this an adaptability ratio that we consider might be related to some type of motor learning.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be able to stand with their eyes closed for 30 seconds without falling

Exclusion Criteria:

* All subjects who are not able to stand with their eyes closed for 30 seconds without falling

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects will be accepted from participants who are over the age of 50 years at the September, 2008 AARP convention in Washington, DC. All subjects must be able to stand with their eyes closed for 30 seconds without falling to be considered eligible for the research study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Forceplate dynamic posturography test | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Study Chair — Carrick Institute for Graduate Studies
Locations (1):
- Walter E. Washington Convention Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No